CLINICAL TRIAL: NCT06681402
Title: Phase I Single-blind Clinical Trial to Evaluate the Safety and Local Immune Activation of a Toll-like Receptor 5 Agonist (FLAMOD) Administered by Aerosol
Acronym: NEBUFLAG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C20-48; 2024-515933-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pneumonia
Keywords: Immunotherapy; Inhalation; Antibiotic resistance; Flagellin; Pneumonia
MeSH Terms: conditions — Pneumonia; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLAMOD (Experimental)
  Interventions: Drug: FLAMOD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FLAMOD — FLAMOD (GMP-grade flagellin) inhalation
  Arms: FLAMOD
Drug: Placebo — Placebo inhalation
  Arms: Placebo

SUMMARY:
This is a single-blind, randomized, placebo-controlled, dose-escalation phase I monocentric trial assessing a single administration of FLAMOD by aerosol in healthy subjects. The recruitment is performed by the Clinical Investigation Center of Tours. This trial is divided in two stages:

* the "start-up phase" consisting of a dose escalation to ensure the safety of FLAMOD while allowing sufficient information on the molecule activity to be accumulated
* the dose-finding phase estimating several dose-activity models and then selecting the one that best fits the data to then propose the dose for the next cohort of participants.

ELIGIBILITY:
Inclusion Criteria:

* provision of signed and dated informed consent form
* stated willingness to comply with all trial procedures, clinic visits, blood draws, and availability for the duration of the trial
* human subjects who are between 18 and 65 years of age
* weight of at least 50 kg and body mass index (BMI) within the range of 18 - 30 kg/m²
* females of non-childbearing potential or of childbearing potential with effective contraception, males willing to practice contraception or having a partner using contraception (if having heterosexual intercourse)
* non-smoker subject (included e-cigarette smoking) since at least 3 months and able to not smoke during the whole trial
* maximum alcohol consumption defined as: i. no more than ten standard glasses per week; ii. no more than two standard glasses per day; iii. having alcohol-free day during the week
* volunteer should be healthy after a clinical examination
* affiliation with a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* febrile and/or suspected infection
* history of chronic pulmonary disease
* history of acute pulmonary disease in the past 6 months
* immunocompromised individuals, which includes immunodeficient patients (e.g., those with asplenism, acquired immune deficiency syndrome, or immunoglobulin deficiencies), patients with haematological diseases or solid cancers, solid organ or stem-cell transplant recipients, as well as patients with other conditions requiring immunosuppression (e.g., rheumatic and autoimmune diseases, inflammatory bowel disease, or multiple sclerosis)
* administration, less than 5 x t1/2 before FLAMOD's administration, of any medication or treatment that may alter the FLAMOD immune responses, such as but not limited to:

  * systemic corticosteroids exceeding 10 mg/day of prednisone equivalent for more than 7 consecutive days or for 10 or more days in total, within 1 month prior to the visit 1. Inhaled and intranasal steroid preparations whatever the dose within 1 month prior to the visit 1.
  * cytotoxic, antineoplastic, immunosuppressant drugs including: calcineurin inhibitors immunoglobulin, mTOR inhibitors, JAK inhibitors, unspecific immunosuppressors, TNF-alpha inhibitors, immunosuppressive monoclonal antibodies [e.g., rituximab or infliximab], any anti-cytokine biological treatment (e.g. TNF-alpha inhibitors, anti-IL6 agents, anti-IL1 agents); within 12 months prior to the visit 1.
  * concurrent immunostimulant drugs or biologic agents including: growth factors, cytokines, interleukins, interferons; within 12 months prior to the visit 1.
  * administration of vaccine within 1 month prior to visit 1.
* administration of anticoagulant treatments: warfarin (coumadin), fondaparinux, heparin (unfractionated Heparin), low molecular weight heparin (enoxaparin, dalteparin), direct oral anticoagulants (rivaroxaban, apixaban, edoxaban, dabigatran); within 1 week prior to the visit 1
* pregnant or lactating woman
* inability to tolerate a nebulization test with saline
* clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 150 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm)
* abnormal ECG that is, in the investigator's opinion, clinically significant including: heart rate <50 BPM, PR interval > 220 ms, QRS interval ≥ 120 ms, QTc interval > 450 ms (QT corrected using Bazett's method), second or third-degree atrioventricular block, any rhythm, other than sinus rhythm, that is interpreted by the investigator to be clinically significant
* subjects whose baseline laboratory values are outside of the normal range, as shown in Appendix 3 - Normal laboratory values unless the abnormality is considered not to be of clinical relevance by the investigator
* positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests
* positive urine nicotine test
* positive urine multi-drug test
* abnormal chest x-ray
* clinically significant abnormality of baseline spirometry tests: forced vital capacity (FVC) <90% predicted; forced expiratory volume in one second (FEV1) <80% predicted; FEV1/FVC ratio <80% or diffusion capacity of the lung for carbon monoxide (DLCO) <70% predicted
* history or presence of drug or chronic alcohol abuse
* history of severe psychiatric disorders that may affect participation in the trial
* significant concurrent illness and any other condition that, in the opinion of the investigator, would compromise the safety or rights of a volunteer participating in the trial or render the subject unable to comply with the protocol
* person subject to a legal protection measure
* subject in the exclusion period of a previous study
* known allergy or intolerance to study drug (including any of its constituents, e.g. FLAMOD and polysorbate 80)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a single administration dose of FLAMOD | From enrollment to the end of follow-up (at 2 weeks +/- 4 days post administration)
  The safety of FLAMOD is assessed via the proportion of Serious Adverse Events, critical safety events, serious adverse reactions, and cytokine release syndrome grade 2 and above.
  The tolerability of FLAMOD is assessed via the proportion of treated participants who experience laboratory abnormalities and/or Adverse Events as defined by Common Terminology Criteria for Adverse Events v5.0.

SECONDARY OUTCOMES:
FLAMOD immune activating dose (IAD) | From enrollment to visit 2 (24 hours + 3-day window post administration)
  Biological activity of FLAMOD is assessed by systemic biomarker surrogates. The lowest dose that reaches immune activation in a maximum number of healthy volunteers is considered as IAD.
Local immune-enhancing effect of FLAMOD on nasal epithelial lining fluid | From enrollment to visit 2 (24 hours + 3-day window post administration)
  Multiomic analyses (proteomic and transcriptomic analyses) will be performed subsequently on nasal epithelial lining fluid collected by nasosorption for proteomic study with a special focus on IL-6, IL-8, CCL20 but not only.
Local immune-enhancing effect of FLAMOD on nasal epithelial cells | From enrollment to visit 2 (24 hours + 3-day window post administration)
  Multiomic analyses (proteomic and transcriptomic analyses) will be performed subsequently on nasal epithelial cells collected by nasal curettage for transcriptomic study to identify differentially expressed genes and pathways.
Systemic immune-enhancing effect of FLAMOD | From enrollment to visit 2 (24 hours + 3-day window post administration)
  Multiomic analyses (proteomic and transcriptomic analyses) will be performed subsequently on blood collected for proteomic study to complete the characterization of the immune response, in addition to IL-6, CRP, PCT and neutrophils that will be available in blood in a short turnaround time.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Guillon, MD, Principal Investigator — Centre Hospitalier Régional Universitaire de Tours
Locations (1):
- Centre hospitalier régional universitaire de de Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
Data and/or samples obtained through this study may be provided to perform new researches on immunology and infectiology fields. Data or samples shared will be coded. The request will be assessed by the sponsor with scientific advice and may require agreement (e.g. a data/material transfer agreement) and accomplishment of regulatory process (e.g. competent authority authorisation) before sharing of data and/or samples with the requesting party.